CLINICAL TRIAL: NCT03299972
Title: Effects of 12 Weeks Resistance Exercise and Whey Protein Supplementation on Energy Metabolism, Appetite, Body Composition and Biomarkers Related to Sarcopenia and Metabolic Health
Brief Title: Multidisciplinary Research Into the Effects of Resistance Exercise and Whey Protein Supplementation in Healthy Older Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coventry University (Other)
Collaborators: University Hospitals Coventry and Warwickshire NHS Trust (Other)
Responsible Party: Principal Investigator, Corbin Griffen, Principle Investigator, Coventry University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: P59723
Record Dates: First submitted 2017-09-11; First posted 2017-10-03 (Actual); Last update posted 2019-07-26 (Actual); Status verified 2019-07

CONDITIONS: Sarcopenia; Muscle Atrophy
Keywords: Sarcopenia; Resistance exercise; Protein
MeSH Terms: conditions — Sarcopenia; Muscular Atrophy | interventions — Whey Proteins; Resistance Training

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Control (Placebo Comparator)
  Interventions: Dietary Supplement: Control
- Whey Protein (Experimental)
  Interventions: Dietary Supplement: Whey Protein
- Resistance Exercise + Control (Experimental)
  Interventions: Dietary Supplement: Control; Other: Resistance Exercise
- Resistance Exercise + Whey Protein (Experimental)
  Interventions: Dietary Supplement: Whey Protein; Other: Resistance Exercise

INTERVENTIONS:
Dietary Supplement: Whey Protein — 25 g whey protein supplementation twice daily (breakfast and lunch)
  Arms: Resistance Exercise + Whey Protein; Whey Protein
Dietary Supplement: Control — 23.75 g maltodextrin twice daily (breakfast and lunch)
  Arms: Control; Resistance Exercise + Control
Other: Resistance Exercise — 60 minutes of resistance exercise twice a week
  Arms: Resistance Exercise + Control; Resistance Exercise + Whey Protein

SUMMARY:
The aim of this randomised, double-blind, placebo-controlled, parallel groups trial is to investigate the effects of 12 weeks resistance exercise and whey protein supplementation on energy metabolism, markers of appetite, inflammation and hormonal response and body composition and strength and functional performance.

Generally healthy, retired men aged 60-80 years will be recruited (n = 52 in total, n = 13 per group). Participants will be randomised to either: a) control group, b) whey protein supplement group, c) resistance exercise + control group or d) resistance exercise + whey protein supplementation group.

DETAILED DESCRIPTION:
With demographics indicating that the world's population aged >60 years will increase from 600 million reported in 2000, to >2 billion by 2050, there is an increasing interest in health issues related to ageing. One area of particular interest is sarcopenia, defined as the progressive loss of muscle mass, strength and physical function as a consequence of ageing. Sarcopenia has been associated with an increase in cardiovascular disease, poor metabolic and cognitive function, reduced quality of life and early mortality. Studies have reported beneficial effects of both resistance exercise and increasing protein intake independently and in combination on markers of sarcopenia (mostly increases in muscle mass, strength and physical function). However, little is known about the effects of combined intervention on energy metabolism, appetite and cognitive and endocrine function. This randomised, double-blind, placebo-controlled, parallel groups trial will investigate these, alongside assessing the effects of combined intervention on total lean tissue mass, muscular strength and functional performance.

ELIGIBILITY:
Inclusion Criteria:

* Retired Men aged 60-80 years
* Body Mass Index 18.5-30 kg/m2
* Not participated in resistance exercise within the last 6 months
* Free from musculoskeletal injury

Exclusion Criteria:

* Retired Men aged <60 or >80 years
* Current smokers, or ex-smokers ceasing <6 months ago
* Body Mass Index <18.5 and >30 kg/m2
* Currently participating in resistance exercise regularly (within last 6 months)
* Not weight stable and/or looking to start a weight loss programme
* Individuals participating in another research project (within the last 6 months) involving dietary and/or exercise intervention
* Existing or past medical history of vascular disease, cancer, diabetes, neurological, kidney, pulmonary, digestive (Coeliac disease), thyroidal disease, osteoporosis or history of falls
* Currently taking protein/amino acid supplements regularly
* Currently prescribed non-steroidal anti-inflammatory medication, hormone replacement therapy (HRT), diabetic medication, beta-blockers, statins
* Uncontrolled blood pressure (Blood pressure >160/100 mmHg)
* Self-reported lactose intolerant or allergic to wheat or potatoes
* Individuals with a pacemaker
* Neuromuscular disorders or injuries

Ages: 60 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2017-10-27 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Changes in components of 24-h energy expenditure and its components (kcal/d) | 0 to 12 weeks
  Measured by whole-room calorimetry
Changes in body composition (kg) | 0 to 12 weeks
  Fat-free mass, fat mass, skeletal muscle mass measured by bio-electrical impedance analysis
Changes in 24-h substrate oxidation (g/d) | 0 to 12 weeks
  Measured by whole-room calorimetry

SECONDARY OUTCOMES:
Biochemical: Appetite hormones | 0 to 12 weeks
  Ghrelin, leptin, and PYY
Biochemical: Insulin Resistance (HOMAR-IR) | 0 to 12 weeks
Salivary:Diurnal Cortisol | 0 to 12 weeks
Biochemical: Inflammtion | 0 to 12 weeks
  Tumor necrosis factor alpha (TNF-α), C-reactive protein (CRP), interleukin-6 (IL-6), interleukin-10 (IL-10), Annexin A1
Interstitial Glucose | 0 to 12 weeks
  24 Hour Continuous Glucose Monitoring
Biochemical: Insulin-Like Growth Factor 1 (IGF-1) | 0 to 12 weeks
Isotonic Strength (kg) - Leg press and leg extension | 0 to 12 weeks
Short Physical Performance Battery (SPPB) | 0 to 12 weeks
  Balance, Gait speed and time to sit and stand from a chair 5 times
Cognitive Function - Cambridge Cognition Neuropsychological Testing Battery | 0 to 12 weeks
Handgrip strength (kg) | 0 to 12 weeks
Biochemical: Myostatin | 0 to 12 weeks
Habitual Physical Activity | 0 to 12 weeks
  Accelerometer
Endurance (Six Minute Walk Test) | 0 to 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Derek Renshaw, PhD, Study Director — Coventry University; John Hattersley, PhD, Study Director — University Hosptials Coventry and Warwickshire NHS Trust; Michael Duncan, PhD, Study Director — Coventry University; Corbin Griffen, MSc, Principal Investigator — Coventry University
Locations (1):
- Coventry University, Coventry, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Griffen C, Renshaw D, Duncan M, Weickert MO, Hattersley J. Changes in 24-h energy expenditure, substrate oxidation, and body composition following resistance exercise and a high protein diet via whey protein supplementation in healthy older men. Physiol Rep. 2022 Jun;10(11):e15268. doi: 10.14814/phy2.15268. PMID 37815091
- [Derived] Griffen C, Duncan M, Hattersley J, Weickert MO, Dallaway A, Renshaw D. Effects of resistance exercise and whey protein supplementation on skeletal muscle strength, mass, physical function, and hormonal and inflammatory biomarkers in healthy active older men: a randomised, double-blind, placebo-controlled trial. Exp Gerontol. 2022 Feb;158:111651. doi: 10.1016/j.exger.2021.111651. Epub 2021 Dec 9. PMID 34896568